CLINICAL TRIAL: NCT01742000
Title: Double-blinded Placebo-controlled Study of Anti-atherosclerotic Activity of Karinat in Postmenopausal Women
Brief Title: Study of Anti-atherosclerotic Activity of Karinat in Postmenopausal Women
Acronym: PEARS-POST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAR-KT-POST
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-09

CONDITIONS: Atherosclerosis
Keywords: postmenopause; phytoestrogen; atherosclerosis; intima-media thickness
MeSH Terms: conditions — Atherosclerosis | interventions — karinat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Karinat (Active Comparator): Karinat 500 mg tablet by mouth three times a day
  Interventions: Dietary Supplement: Karinat
- Sugar pill (Placebo Comparator): Placebo 500 mg tablet by mouth three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Karinat
  Arms: Karinat
Drug: Placebo — Sugar pill manufactured to mimic Karinat 500 mg tablet
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to investigate the anti-atherosclerotic action of natural drug Karinat based on phytoestrogen-rich botanicals in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 5 years after menopause
* Maximum intima-media thickness of common carotid artery more than 0,80 mm (ultrasonographic B-mode examination)
* The absence of climacteric syndrome (less than 3 points by Blatt-Kupperman scale)
* The absence of chronic diseases demanding permanent drug administration (more than 2 month per year)
* The absence of hypolipidemic therapy or hormone replacement therapy during 6 months before the inclusion

Exclusion Criteria:

* Administration of lipid-lowering drugs, and/or hormone replacement therapy, and/or phytoestrogens during 6 month before inclusion
* Continuous administration of sulfonylurea derivatives, and/or beta-blockers, and/or calcium antagonists (more than 2 months per year)
* Personal history or diagnostic of following diseases:

  1. Personal history of stroke, coronary heart disease, acute myocardial infarction or transient ischemic attacks
  2. Pulmonary thromboembolism
  3. Chronic heart failure IIa-III
  4. Uncontrolled arterial hypertension (systolic blood pressure > 145 mmHg, diastolic blood pressure > 95 mmHg under hypotensive therapy)
  5. Malignancy
  6. Chronic renal failure II-III
  7. Chronic hepatic failure II-III
  8. Liver cirrhosis
  9. Individual intolerance of Karinat or major side effects

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
B-mode ultrasound of carotid arteries | up to 2 years
  Variation of intima-media thickness of common carotid arteries

SECONDARY OUTCOMES:
Measure of serum atherogenicity | up to 2 years
  Change of the ability of serum to induce cholesterol accumulation in cultured cells